CLINICAL TRIAL: NCT06454552
Title: A Study of Stimulant Medications Infusion Through Midline Catheters Based on Real-world Data
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-2082-01
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Catheter Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- irritant medications group: Patients who used midline catheter to infuse irritant medications.
- nonirritant medications group: Patients who used midline catheter to infuse nonirritant medications.

SUMMARY:
Based on the previous research, this study intends to explore the outcome of trans-MC infusion of stimulant drugs when the MC tip is located in the subclavian vein/chest wall segment axillary vein, especially to analyze the relationship between drug dose, infusion days and catheter-related complications, so as to provide a basis for the clinical application of MC infusion stimulant drugs, provide evidence for the revision of infusion practice guidelines, and ensure the safety of patients' infusion. Reduce the occurrence of adverse events, provide a basis for further expanding the clinical application scope of MC, reduce unnecessary peripherally inserted central venous catheters (PICC) and central venous catheters (CVC) and other central venous catheters, and reduce medical costs.

DETAILED DESCRIPTION:
Midline catheters were inserted by hospital nurses in each center, and patients with MC catheters were included in order, and baseline data of patients were extracted from medical records, including patients' age, gender, education level, body mass index, occupation, admission diagnosis, thrombosis history, major surgery trauma history, chronic medical history, catheterization history and related examination indicators. At the same time, researchers authorized by the principal investigators of each center and uniformly trained researchers will collect data and record the puncture situation during catheterization: including catheter, puncture method, puncture location, puncture arm, puncture site, punctured blood vessel and vascular diameter, number of puncture needles, catheter brand, catheter model, catheter insertion length, catheter exposed length, catheter tip position; During the catheter indwelling period, the catheter function and complications were collected until extubation, and the reasons for extubation, transcatheter blood collection, and vascular intima were recorded, and the patient's transcatheter drug information was extracted from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old.
* In patients with conventional indwelling single-chamber three-way valve MC, the catheter tip is located in the axillary vein or subclavian vein of the chest wall segment.

Exclusion Criteria:

* Those who have been placed with a central venous catheter during MC insertion.
* Vulnerable groups, including people with mental illness, cognitive impairment, critically ill patients, minors, pregnant women, illiterates, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study intends to prospectively include patients who have been admitted to multiple centers such as Sir Run Run Shaw Hospital (team leader unit) affiliated to Zhejiang University School of Medicine and have MC implanted.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-06-11 (Estimated); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
catheter complications | during catheter indwelling procedure
  catheter complications rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Linfang, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao L, Cao X, Liu C, Wang J, Jin X, Zeng X, Li X, Zhuang Y. Impact of irritating infusates via midline catheters on vascular complications: a multicentre prospective cohort study protocol in China. BMJ Open. 2025 Aug 31;15(8):e093180. doi: 10.1136/bmjopen-2024-093180. PMID 40887123